CLINICAL TRIAL: NCT06037928
Title: Plasma Sodium and Sodium Administration in the ICU. A Retrospective Observational Study.
Brief Title: Plasma Sodium and Sodium Administration in the ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Hans Bahlmann, Sponsor, University Hospital, Linkoeping
Other Study IDs: IVA-salt
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Hypernatremia; Hyponatremia; Critical Illness
Keywords: Fluid Therapy; ICU; Drug Prescription
MeSH Terms: conditions — Hypernatremia; Hyponatremia; Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients in the Intensive Care Unit often present with low levels of plasma sodium and are therefore often administered high amounts of sodium, both as an additive to intravenous glucose solutions and as a constituent of various drugs and infusion fluids. Recent findings question the benefit of these large quantities of sodium and raise the question whether the individual physician takes the total sodium administration into account when sodium additives are prescribed. It can also be suspected that sodium prescription differs significantly between physicians.

DETAILED DESCRIPTION:
Treatment with intravenous fluids (fluid therapy) is a cornerstone in intensive care. The primary aim of fluid therapy is to optimize the amount of fluid in the various spaces of the body: intravascularly (plasma), intracellularly and interstitially. Secondarily, one tries to optimize the constitution of fluid in plasma, since this is the only fluid space that is available for analysis. Fluid constitution is referring to the physical properties such as pH-value, osmolality, and partly the concentration of different elements solved in plasma (i.e. sodium, potassium, chloride, magnesium, and proteins like albumin). For this reason, there are a lot of different fluids that the physician in the intensive care can choose from. In addition, the physician can also choose to prescribe different additives to adapt these fluids to fulfil the individual patient's needs. Therefore, to prescribe both the amount and constituency of fluid therapy is a key task for ICU-physicians.

One of the most important additives to be prescribed is sodium. Sodium is the molecule (except for water) that has the highest concentration in plasma (normally around 140 mmol/L) and is therefore of utmost importance for plasma osmolality. Sodium concentration in plasma is often decreased in critically ill patients (hyponatremia) which, in turn, is associated with a worse outcome, and thus a normal task for an ICU-physician to attempt to regulate through administering amounts of sodium that are substantially higher than the physiological needs.

Recent findings have revealed that there is a large variation between different physicians when it comes to the amount of fluid the patient receives, a variation that has no scientific basis.

Fluids used in the operating room and in the intensive care often contain large quantities of sodium to create a physiological osmolality. It is thus hypothesized that it is not only the large quantities of fluid that causes a worse outcome in fluid overload, but also the un-physiologically large amount of administered sodium.

The aim of the study is partly to gain knowledge about how sodium prescription is performed in clinical practice in the intensive care, as well as how this administration relates to actual changes in plasma sodium.

Statistical method: Normal distribution will be tested via the Shapiro-Wilks test. All tests of significance are performed two-sided. P-value lower than 0.05 is considered significant. No corrections for multiple comparisons are performed if nothing else is stated.

Missing values: Single missing values are principally not replaced. In exceptional cases, if missing data leads to a whole series of data being misleading, then missing data can be imputed by calculating the mean of two adjacent values, under the condition that this results in a reasonable value.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Documented length of stay at the Central Intensive Care Unit (CIVA) at the University Hospital of Linköping of seven (7) days minimum.
* The patient has been discharged from the ICU.
* Body Mass Index (BMI) between 18.0 and 48.0 kg/m2 at admission.

Exclusion Criteria:

* The patient has previously been included in the study in connection with another ICU-admission.
* The patient has a severe hyponatremia (<129 mmol/L) upon arrival to the ICU.
* The patient has a severe hypernatremia (>149 mmol/L) upon arrival to the ICU.
* The patient is severely hyperosmolar (>330 mmol/L) upon arrival to the ICU.
* The patient is severely hyperglycemic (>30 mmol/L) upon arrival to the ICU.
* The patient has an elevated serum urea (>30 mmol/L) upon arrival to the ICU.
* The patient receives any dialysis treatment during the observation time.
* The patient is suspected to have an elevated intracranial pressure during the observation time or is suspected to have other intracranial pathology that is likely to affect sodium homeostasis
* The patient has an intoxication with toxic alcohols as a primary diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with a documented length of stay at the Intensive Care Unit of seven days minimum
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
The coefficient of determination (r2) between the amount prescribed sodium additive and the amount of sodium the patient is expected to receive through other routes. | During admission to ICU for a maximum of 28 days
  The amount of sodium additive is defined as the amount of sodium in mmol/kg ABW (actual body weight) that is being given in glucose solutions during the coming 24 hours.
  Example: A patient weighing 70 kilograms is being prescribed intravenous glucose of 1L, with an additive of 40 mmol of sodium during 12 hours. The amount of additive will then be calculated as (40+40)×2⁄70=2.3 mmol/kg
  The amount of expected sodium administrated, per kg and day, is defined as the sodium contents of:
  1. Enteral and/or parenteral nutrition during one day.
  2. Drugs administered through infusion pumps during one day.
  3. Other fluids that have been prescribed during the morning round.

SECONDARY OUTCOMES:
The coefficient of determination (r2) in a multivariate analysis where prescribing physician is the independent variable and the amount of prescribed sodium additive is the dependent variable. | During admission to ICU for a maximum of 28 days
  Only data points where administering physician has been registered and where plasma sodium is < 150 mmol/L are included. Data will, however, be displayed for all levels of plasma sodium. The amount of sodium additive is defined as the amount of sodium in mmol/kg ABW that is prescribed through glucose infusion the coming day.
Difference in median or mean in the amount of prescribed sodium additive between anesthesiologists mainly working in intensive care, anesthesiologists mainly working with patients undergoing surgery and between resident physicians. | During admission to ICU for a maximum of 28 days
  Only data points where administering physician has been registered and where plasma sodium is < 150 mmol/L are included. Data will, however, be displayed for all levels of plasma sodium. Information regarding chief working area will be retrieved through the schedule of the clinic.
Difference in median or mean in the amount of prescribed sodium additive between physicians born no later than 12-31-1982 and physicians born 1983 and later. | During admission to ICU for a maximum of 28 days
  Only data points where administering physician has been registered and where plasma sodium is < 150 mmol/L are included. Data will, however, be displayed for all levels of plasma sodium. Information regarding birth year is retrieved through an official database (www.mrkoll.se).
The coefficient of determination (r2) between plasma sodium and the amount of prescribed sodium additive. | During admission to ICU for a maximum of 28 days
  Only data points where plasma sodium is < 150 mmol/L are included. Data will, however, be displayed for all levels of plasma sodium.
The coefficient of determination (r2) between the amount of prescribed sodium additive and observed changes in plasma sodium. | During admission to ICU for a maximum of 28 days
  Calculated in intervals of 1, 2, 3, 4 and 5 days
The coefficient of determination (r2) between the total amount of administered sodium and observed changes in plasma sodium. | During admission to ICU for a maximum of 28 days
  Calculated in intervals of 1, 2, 3, 4 and 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Linköping, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Carvalho H, Letellier T, Karakachoff M, Desvaux G, Caillon H, Papuchon E, Bentoumi-Loaec M, Benaouicha N, Canet E, Chapelet G, Le Turnier P, Montassier E, Rouhani A, Goffinet N, Figueres L. Hyponatremia is associated with poor outcome in COVID-19. J Nephrol. 2021 Aug;34(4):991-998. doi: 10.1007/s40620-021-01036-8. Epub 2021 Apr 7. PMID 33826113
- [Background] Lilot M, Ehrenfeld JM, Lee C, Harrington B, Cannesson M, Rinehart J. Variability in practice and factors predictive of total crystalloid administration during abdominal surgery: retrospective two-centre analysis. Br J Anaesth. 2015 May;114(5):767-76. doi: 10.1093/bja/aeu452. Epub 2015 Jan 13. PMID 25586725
- [Background] Van Regenmortel N, Moers L, Langer T, Roelant E, De Weerdt T, Caironi P, Malbrain MLNG, Elbers P, Van den Wyngaert T, Jorens PG. Fluid-induced harm in the hospital: look beyond volume and start considering sodium. From physiology towards recommendations for daily practice in hospitalized adults. Ann Intensive Care. 2021 May 17;11(1):79. doi: 10.1186/s13613-021-00851-3. PMID 33999276